CLINICAL TRIAL: NCT04387149
Title: Biomarkers of Acute Kidney Injury Following Cardiopulmonary Bypass Surgery-supported Cardiac Surgery
Brief Title: Biomarkers of Acute Kidney Injury Following Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Erick McNair, Research Scientist, University of Saskatchewan
Other Study IDs: Bio 113
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Novel Biomarkers of Acute Kidney Injury Following Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CSA-AKI: Patients that developed cardiac surgery-associated Acute Kidney Injury
- non CSA-AKI: Patients that did not developed cardiac surgery-associated Acute Kidney Injury

SUMMARY:
Acute kidney injury occurs in up to 30% of patients undergoing cardiac surgery. Cardiac surgery associated-acute kidney injury (CSA-AKI) is characterized by a sudden and sustained decrease in renal function with insufficient elimination waste products. The problem is that postoperative diagnosis of CSA-AKI is delayed because it relies solely upon the slow and unreliable rise in serum creatinine (SCr) levels that may lead to delayed start in treatment and increased risk of adverse outcomes. We hypothesize that Matrix Metalloproteins (MMPs) -2, -9 and Neutrophil gelatinase-associated lipocalin (NGAL) are associated with and earlier detectors of CSA-AKI compared to levels of SCr.

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB), although essential to the performance of most cardiac operations, has been shown to cause injury to other organs, particularly to the kidneys and brain. Matrix Metalloproteins (MMPs) are ubiquitous proteolytic enzymes that degrade extracellular matrix and have been shown to be involved in injury to transplant kidneys. To date, no interventions are available to decrease the risk of cardiac surgery associated-acute kidney injury (CSA-AKI).

NGAL is a known indicator of injury to kidney, thus making it a promising biomarker for CSA-AKI. It may be that a single biomarker will not be sensitive and specific across the spectrum of CSA-AKI. This research investigates MMP-2, -9 and Neutrophil gelatinase-associated lipocalin (NGAL) and their association with and earlier detection of CSA-AKI compared to levels of SCr.

We hypothesize that increased activity of MMPs are associated with CSA-AKI. Furthermore, MMP-2 and/ or -9 may be predictors and/ or biomarkers for the early detection of CSA-AKI compared to serum levels of creatinine.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria consisted of both sexes, 18-85 years of age, undergoing elective or urgent cardiac surgery with a hemoglobin (Hgb) >100 g/L.

Exclusion Criteria:

* The exclusion criteria included were patients for emergent surgery, pre-existing chronic kidney disease (eGFR<30 mL/min) on dialysis or prescribed nephrotoxic mediations.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Approached as a prospective study male and female patients undergoing cardiopulmonary bypass-supported cardiac surgery were recruited and signed a written consent agreeing to participate in this research.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Increased MMP-2 and -9 in patients that develop CSA-AKI | Pre-CPB, 10 min post-CPB time point, 4 hours post-CPD
  Increased MMP-2 and -9 activity in serum and or urine in patients that develop CSA-AKI

SECONDARY OUTCOMES:
Increased NGAL levels in patients that develop CSA-AKI | Pre-CPB, 10 min post-CPB time point, 4 hours post-CPD
  Increased NGAL levels in serum and or urine in patients that develop CSA-AKI

CONTACTS AND LOCATIONS:
Overall Officials: Erick D McNair, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Undecided